CLINICAL TRIAL: NCT01539187
Title: Symptom Effectiveness Study of VizAblate® Intrauterine Ultrasound-Guided RF Ablation (IUUSgRFA) in the Ablation of Large Uterine Fibroids
Brief Title: Fibroid Ablation Study - Large Fibroids
Acronym: FAST-L
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Investigational device changes
Sponsor: Gynesonics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CL 03536
Record Dates: First submitted 2012-02-21; First posted 2012-02-27 (Estimated); Last update posted 2015-03-17 (Estimated); Status verified 2015-03

CONDITIONS: Leiomyoma; Uterine Fibroids; Menorrhagia
Keywords: uterine fibroid RF ablation; intrauterine ultrasound; VizAblate
MeSH Terms: conditions — Leiomyoma; Menorrhagia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- VizAblate intervention (Experimental): VizAblate System with subject serving as her own control
  Interventions: Device: VizAblate System

INTERVENTIONS:
Device: VizAblate System — VizAblate enables a minimally invasive procedure to visualize, target, and ablate uterine fibroids using intrauterine ultrasound and radiofrequency (RF) energy

SUMMARY:
The purpose of this study is to establish the effectiveness and confirm the safety of the VizAblate System in the ablation of large (> 5 cm) symptomatic uterine fibroids.

ELIGIBILITY:
Inclusion Criteria:

* 28 years of age or older
* Consistent menstrual cycles
* History of excessive bleeding for at least 3 months
* Baseline UFS-QOL Symptom severity score ≥ 20
* At least one target fibroid having a maximum diameter > 5cm and ≤ 10 cm
* Not at material risk for pregnancy
* Willingness to participate, adhere to follow-up requirements, and sign the informed consent form
* Willing to have uniform maintenance of antifibrinolytic or non steroidal anti-inflammatory agents
* Menstrual Pictogram score ≥ 120 during a one-month screening period.

Exclusion Criteria:

* Presence of type 0 intracavitary fibroids
* Target fibroid > 10cm in maximum diameter
* Abnormality of the endometrial cavity that obstructs access of the treatment device
* Postmenopausal
* Desire for current or future fertility
* Hemoglobin < 6 g/dl
* Evidence of disorders of hemostasis
* Use of GnRH agonist or depomedroxyprogesterone acetate or other implantable or injectable progestin and/or estrogen, SERM or SPRM within the last 6 months prior to screening
* Evidence for current cervical dysplasia (CIN II or greater)
* Endometrial hyperplasia
* Confirmed abdominal / pelvic malignancy within previous five years
* Active pelvic infection or positive screen for pelvic gonorrhea or chlamydia
* Clinically significant adenomyosis
* Previous uterine artery embolization
* Previous surgical or ablative treatment for fibroids or menorrhagia within 12 months prior to screening
* Current use of anticoagulant therapy
* Major medical or psychiatric illness affecting general health or ability to adhere to follow-up
* Contraindication to MRI
* Renal insufficiency
* Uncontrolled hypertension lasting 2 years or more
* Calcified fibroids
* Presence of extrauterine pelvic mass
* Presence of tubal implant for sterilization
* Previous pelvic irradiation
* Endometrial cavity length < 4.5 cm

Min Age: 28 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2012-06; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Mean percentage change in target fibroid perfused volume | Baseline, 3 months, 12 months

SECONDARY OUTCOMES:
Number of adverse events | Procedure through 12 mo
  Procedure safety will be assessed by recording all adverse events that occur on the day of the procedure. Longer-term safety will be assessed by recording at each follow-up visit any untoward medical occurrence since baseline. Each adverse event will be assessed for severity and relationship to study device.
Percentage reduction in Symptom Severity Score (SSS) subscale of the Uterine Fibroid Symptom and Quality-of-Life (UFS-QOL) Questionnaire | Baseline through 12 months
Rate of surgical reintervention for menorrhagia | through 12 months
Return to normal daily activity | 2 weeks or until returned to normal activity
Percentage reduction in Menstrual Pictogram score | through 12 months

CONTACTS AND LOCATIONS:
Overall Officials: David Toub, MD, Study Director — Gynesonics
Locations (10):
- Universidad Autonoma de Nuevo Leon (UANL), Monterrey, Nuevo León, Mexico
- Netherlands (4):
  - Maxima Medisch Centrum, Veldhoven, North Brabant
  - Vrije Universiteit Medisch Centrum, Amsterdam, North Holland
  - Medisch Spectrum Twente, Enschede, Overijssel
  - St. Antonius Ziekenhuis, Nieuwegein, Utrecht
- United Kingdom (5):
  - University College Hospital, London, London
  - Royal London Hospital, Whitechapel, London
  - Birmingham Women's NHS Foundation Trust, Birmingham, West Midlands
  - Princess Royal Hospital, Haywards Heath, West Sussex
  - Bradford Teaching Hospitals NHS Trust, Bradford, West Yorkshire